CLINICAL TRIAL: NCT06961227
Title: Comparative Analysis of Ventilation Distribution in Intensive Care: Mandatory Minute Ventilation Versus Synchronized Intermittent Mandatory Ventilation Using Electrical Impedance Tomography"
Brief Title: Effectiveness of Ventilation Modes in Intensive Care: A Comparison of Mandatory Minute Ventilation and Synchronized Intermittant Mandatory Ventilation Using Bioelectrical Impedance Tomography
Status: Recruiting | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Melahat Yalcin Solak, Lecturer Doctor, Harran University
Other Study IDs: HRÜ.24.20.35
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Ventilation Modes; Mechanical Ventilation; Critical Illness; Respiratory Support; Intensive Care Unit (ICU) Patients; Mechanical Ventilation Dependence; Evaluation of Mechanical Ventilation Modes (SIMV and MMV) in Adult Intensive Care Unit Patients Using Electrical Impedance Tomography
Keywords: Mechanical Ventilation; SIMV; MMV; Electrical Impedance Tomography; EIT; Intensive Care Unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patients: Hemodynamically stable adult patients (≥18 years) in the intensive care unit who are receiving mechanical ventilation and are eligible to undergo both SIMV and MMV ventilation modes in a crossover observational design. Patients will be monitored using Electrical Impedance Tomography (EIT) under each mode.
  Interventions: Other: No investigational intervention

INTERVENTIONS:
Other: No investigational intervention — No investigational intervention. Patients will be observed under standard ventilation modes (SIMV and MMV) as part of routine care.

SUMMARY:
Synchronized Intermittent Mandatory Ventilation (SIMV) is a commonly used ventilatory mode available in many modern ventilators, frequently applied in intensive care units for patients requiring invasive mechanical ventilation. SIMV delivers a preset tidal volume or pressure at a predetermined respiratory rate and synchronizes with the patient's spontaneous breathing efforts, thereby enhancing patient-ventilator interaction and contributing to rehabilitation.

Mandatory Minute Ventilation (MMV) is a hybrid mode combining features of SIMV and Pressure Support Ventilation (PSV), guaranteeing a preset minute ventilation (tidal volume × respiratory rate). It synchronizes support based on the patient's spontaneous efforts and compensates in cases of insufficient minute ventilation.

Electrical Impedance Tomography (EIT) is a non-invasive, radiation-free imaging technique that enables real-time monitoring of pulmonary ventilation and perfusion by applying alternating electrical currents through surface electrodes. EIT has demonstrated strong correlation with findings from computed tomography, nitrogen washout, PET, and SPECT imaging modalities.

This study aims to evaluate the effectiveness of MMV compared to SIMV in mechanically ventilated, hemodynamically stable adult patients (>18 years old) in the intensive care unit. Patients must not require vasopressors, have a FiO₂ ≤ 60%, PEEP ≤ 8 cmH₂O, or receive neuromuscular blocking agents.

Patients will be monitored under both SIMV and MMV modes, separated by a 12-hour interval. To minimize carry-over effects, a one-hour washout period will be implemented before data collection with EIT. Key parameters including PO₂/FiO₂ ratio, PaCO₂, and EtCO₂ will be assessed. The sequence of ventilatory mode application will follow a crossover study design.

DETAILED DESCRIPTION:
Synchronized Intermittent Mandatory Ventilation (SIMV) and Mandatory Minute Ventilation (MMV) are two established modes of mechanical ventilation commonly used in intensive care settings. SIMV delivers a fixed number of breaths with preset tidal volume or pressure, while allowing the patient to breathe spontaneously between mandatory breaths, enhancing patient-ventilator synchrony. MMV combines features of SIMV and Pressure Support Ventilation (PSV), ensuring a target minute ventilation by supplementing spontaneous efforts when necessary.

Electrical Impedance Tomography (EIT) is a non-invasive, radiation-free imaging modality that provides real-time monitoring of regional lung ventilation and perfusion through surface electrodes. EIT has been validated against conventional imaging and monitoring methods including computed tomography, nitrogen washout, PET, and SPECT. It enables continuous bedside evaluation of ventilation distribution, making it particularly useful for guiding mechanical ventilation strategies in critically ill patients.

This prospective, single-center, crossover study aims to evaluate the effectiveness and physiological impact of MMV compared to SIMV in adult ICU patients who are hemodynamically stable but require mechanical ventilation due to various non-neuromuscular reasons. Inclusion criteria require patients to be over 18 years old, not on vasopressor therapy, with FiO₂ ≤ 60%, and without the need for high PEEP (>8 cmH₂O) or neuromuscular blockade.

Each patient will be ventilated with both SIMV and MMV modes for 12 hours each, with the order of modes randomized using a crossover design. To eliminate carry-over effects, a one-hour washout period will be implemented between mode transitions. During each ventilation mode, EIT will be used to assess real-time regional ventilation distribution. Additionally, gas exchange parameters including PO₂/FiO₂ ratio, PaCO₂, and EtCO₂ will be recorded. The primary objective is to determine whether MMV offers comparable or superior ventilation distribution and gas exchange compared to SIMV in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Intubated and receiving invasive mechanical ventilation

Hemodynamically stable (no vasopressor support)

FiO₂ ≤ 60%

PEEP ≤ 8 cmH₂O

Not receiving neuromuscular blocking agents

Able to tolerate switching between SIMV and MMV modes

Exclusion Criteria:

Pregnant or breastfeeding patients

Patients with neuromuscular diseases affecting respiratory drive

Unstable hemodynamics or ongoing need for vasopressors

Patients requiring high PEEP (>8 cmH₂O)

Patients with DNR (do not resuscitate) status

Participation in another interventional study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted to the intensive care unit who are intubated and receiving invasive mechanical ventilation. All participants are hemodynamically stable and not receiving vasopressors, high levels of PEEP, or neuromuscular blockers at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Regional Ventilation Distribution Measured by Electrical Impedance Tomography (EIT) | Within 1 hour after initiation of each ventilation mode (SIMV and MMV)
  Comparison of regional lung ventilation patterns between SIMV and MMV modes in mechanically ventilated ICU patients, assessed by EIT imaging.

SECONDARY OUTCOMES:
PO₂/FiO₂ Ratio (Oxygenation Index) | Measured within 1 hour of each mode (SIMV and MMV)
  Arterial oxygen partial pressure (PaO₂) divided by fraction of inspired oxygen (FiO₂), used to assess oxygenation efficiency under each ventilation mode.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University Faculty of Medicine, Department of Anesthesiology and Reanimation, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the limited sample size and the absence of prior consent for data sharing from participants. The collected data is intended solely for internal analysis within the study team.

REFERENCES:
- [Background] Franchineau G, Jonkman AH, Piquilloud L, Yoshida T, Costa E, Roze H, Camporota L, Piraino T, Spinelli E, Combes A, Alcala GC, Amato M, Mauri T, Frerichs I, Brochard LJ, Schmidt M. Electrical Impedance Tomography to Monitor Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2024 Mar 15;209(6):670-682. doi: 10.1164/rccm.202306-1118CI. PMID 38127779
- [Background] Lobo B, Hermosa C, Abella A, Gordo F. Electrical impedance tomography. Ann Transl Med. 2018 Jan;6(2):26. doi: 10.21037/atm.2017.12.06. PMID 29430443
- [Background] Guthrie SO, Lynn C, Lafleur BJ, Donn SM, Walsh WF. A crossover analysis of mandatory minute ventilation compared to synchronized intermittent mandatory ventilation in neonates. J Perinatol. 2005 Oct;25(10):643-6. doi: 10.1038/sj.jp.7211371. PMID 16079905